CLINICAL TRIAL: NCT00959348
Title: The Effect of Inhaled Corticosteroids on the Risk of Diabetes, Impaired Glucose Tolerance and Characteristics of Glucose Regulation in Adults With Asthma : a Population Based Matched Controlled Study
Brief Title: Effect of Inhaled Steroids on Glucose Regulation in Asthma Patients
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr. HO Chung Man James, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 07-291
Record Dates: First submitted 2009-08-09; First posted 2009-08-14 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Asthma
Keywords: Asthma; Diabetes; Impaired glucose tolerance; Insulin resistance
MeSH Terms: conditions — Asthma; Diabetes Mellitus; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma: Asthma patients on inhaled corticosteroids
- Control: Select matched controls from the general population database of Cardiovascular Risk Factor Prevalence Study 2 (CRISPS2)

SUMMARY:
Inhaled steroid has been the cornerstone in the treatment of asthma, which carries a huge patient population worldwide including Hong Kong. In general, the safety of long-term use of inhaled steroid has been well documented. Yet, long-term users of such treatment carry increased risk of complications like cataract. In particular, the exact association of inhaled steroid use and development of diabetes mellitus is not known, despite a clear causal relationship between oral steroid use and diabetes. Therefore this epidemiology study (based on questionnaire and blood tests) aims to investigate the effect of inhaled corticosteroid on the risk of diabetes, impaired glucose tolerance and insulin resistance in adults with asthma. The impact of this study is expected to affect the current practice of long-term use of inhaled corticosteroid especially among patients with asthma.

DETAILED DESCRIPTION:
Inhaled corticosteroids (ICS) have been shown to have many side effects that are consistent with systemic corticosteroids, suggesting that its systemic absorption can lead to adverse effects in the long term users. ICS can pose a major health impact in the community, especially when its use has become widely accepted as mainstay treatment for asthma and chronic obstructive airway diseases in recent decades.

In 1997, inhaled corticosteroids were shown to increase the risk of nuclear cataracts by 1.5-fold and posterior subcapsular cataracts by 1.9-fold respectively. Besides, high dose ICS use for more than 3 months increased risk of open angle glaucoma with OR 1.44. In 1998, a case control study demonstrated positive association of cataract extraction in elderly ICS users. ICS use of more than 3 years increased cataract by 3-fold in high dose users (> 1mg daily budesonide dipropionate). Whereas low dose use (<1mg daily budesonide dipropionate) for more than 2 years increased cataract by 1.6-fold. Subsequent studies also found increased risk of osteoporosis in long term ICS users.

It has been well known that systemic corticosteroid causes diabetes by inducing insulin resistance. Previous study showed a 2-fold increased risk of diabetes in patients using systemic corticosteroids.

Nevertheless, of the many systemic side effects that are known to inhaled corticosteroids, its effect on the risk of diabetes has not been established yet.

There have also been 2 small scale studies about the effect of ICS on insulin resistance profile, however, the study findings were also inconclusive.

In 1987, a study of 9 subjects, given 4 weeks of inhaled budesonide dipropionate 1mg daily, were shown to have increase in 2-hour peak glucose level in oral glucose tolerance test, and also increased fasting serum insulin concentration, suggesting that ICS use was associated with glucose dysregulation and increase insulin resistance. Subsequently, in 1993, another study of 15 subjects with unstable asthma compared to 15 normal control subjects, a reduction in insulin resistance in patients with uncontrolled asthma was noted upon 1 month of ICS treatment; while the insulin resistance profile became static at 5 and 8 months of therapy. This study suggests that insulin resistance profile is increased in subjects with unstable asthma in relation to the stress induced during exacerbation. ICS can reduce insulin resistance profile by stabilizing asthma control.

In terms of researches relating ICS to diabetes, there are limited studies in the elderly. In 1998, a study showed dose dependent worsening of diabetic control in the diabetic elderly using high dose ICS. However, 2 subsequent case control studies conducted in 2002 failed to demonstrate any association of diabetes in elderly with either current use of ICS or 3 years uses of ICS.

These study results are subjected to confounding by concurrent systemic corticosteroid usage, lack of long term users of ICS, as well as the effect of other competing causes of diabetes (ie. aging and obesity) being so strong in the elderly that the impact of ICS on the risk of diabetes might have been masked in this particular group of patients.

So far, data is lacking in terms of the association between inhaled corticosteroids and diabetes, as well as impaired glucose tolerance - the pre-diabetic condition. Moreover, the profile of glucose regulation and potential hyperinsulinemia in ICS users with normal glucose tolerance is largely unexplored.

As Asians are at increased risk of developing NIDDM, the effect of ICS in inducing diabetes in the Chinese might be more prominent than that for subjects in the western countries. It is of more clinical significance and relevance to study this issue in a Chinese dominant community like Hong Kong.

Therefore, we shall investigate the effect of ICS, trying to understand its impact on the whole disease spectrum of insulin resistance. We shall begin with study on the risk of diabetes, then move on to that of impaired glucose tolerance (IGT) and finally to explore potential hyperinsulinemia in subjects with normal glucose tolerance who have used ICS. We will also put particular emphasis on the younger Chinese population, where the impact of age and obesity is less marked, and therefore, the effect of ICS on the risk of DM/IGT/ hyperinsulinemia can be better manifested and delineated.

About 10% of our population has asthma and of these, 50% are on long term inhaled corticosteroids. While asthma is not known to cause diabetes and hence not a confounder for the association of ICS and DM, we shall therefore target at the adult Chinese asthma patients using ICS as our study subjects, and compare the risk of diabetes/IGT/hyperinsulinemia of this group of patients with that of the general population.

Since diabetes mellitus is a major health problem that is strongly associated with multiple cardiovascular morbidity and mortality, and inhaled corticosteroid being the most commonly prescribed drug in treating chronic airway diseases, knowledge regarding the risk of DM in association with chronic ICS use will be of major impact on public health.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients who have follow-up in our asthma clinics; OR Eligible subjects belonging to 1996 population cohort, which represents the general population ie. same base population as the asthma patients
* Current inhaled corticosteroid users

Exclusion Criteria:

* On maintenance oral steroid
* Oral steroid use within 180 days prior to study
* IDDM
* Known secondary causes for diabetes including pregnancy, cushing's syndrome and acromegaly
* Inhaled corticosteroid use for < 6 months
* Asthma exacerbation in recent 1 month, yet without need for systemic steroid use, as previous study has shown increased insulin resistance in subjects with unstable asthma, in relation to the acute stress during attack, which subsequently returned to normal after 1 month on disease stabilization

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients will be recruited from asthma clinic in Queen Mary Hospital, Queen Elizabeth Hospital, Kowloon Hospital, Kwong Wah Hospital and select matched controls at 1:1 ratio from the general population database of Cardiovascular Risk Factor Prevalence Study 2 (CRISPS2).
Sampling Method: Non-Probability Sample
Enrollment: 1394 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To investigate the ICS effect on the risk of DM/IGT/insulin resistance | 1 year

SECONDARY OUTCOMES:
To study the dose response relationship and effect modifying factors if risk is present | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chung-man James Ho, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Kowloon Hospital, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong